CLINICAL TRIAL: NCT05534932
Title: Guideline-directed Management and Therapy (GDMT) for the Prevention of Postpartum Cardiac Dysfunction in Preeclamptic African American Women
Acronym: GDMT For PE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB 22-1412
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Preeclampsia Postpartum
Keywords: Preeclampsia; Postpartum GLS Levels; Postpartum Activin A Levels; Cardiac Postpartum Therapy; Hypertension; Cardiovascular disease
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized at baseline into one of two arms for the purposes of the sub-study. One arm will receive the GDMP, which includes the RPM program. The other arm will not receive the GDMP and will continue thier usual standard of care course per thier treating physician.
Masking Description: No blinding between arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Arm (Active Comparator): 35 Subjects will be placed in the sub-study treatment arm. These subjects will receive the remote patient monitoring program therapy offered by the University of Chicago heart failure program.
  Interventions: Device: Remote Patient Monitoring
- Observational Arm (No Intervention): 35 Subjects will be placed in the sub-study Obervational arm. These subjects will not reveive the remote patient monitoring program and will continue with thier standard of care treatment for the duration of the study.

INTERVENTIONS:
Device: Remote Patient Monitoring — Subjects in this group will receive RPM therapy through the University of Chicago Heart Failure program. This therapy consist of a bluetooth tablet, blood pressure cuff and a health scale for subjects to bring home and take thier measurements on a daily bases up to their 3 month clinic visit. This data will then be transmitted to EPIC where the study team will retrieve the data.
  Other Names: RPM
  Arms: Treatment Arm

SUMMARY:
This is a single-center, open-label pilot study looking at how Guideline-directed management and therapy (GDMP) in post-partum women with preeclampsia can improve Global Longitudinal Strain (GLS).

DETAILED DESCRIPTION:
This study is looking at when given GDMP in post-partum women with preeclampsia, compared to the current standard of care, can this therapy improve Global Longitudinal Strain (GLS) at 9 months. Subjects who agree to participate and who have already completed the PARENT study (NCT04479072) at 6-months will be randomized in this study to either the GDMP (Treatment) arm or the standard of care (Observational) arm. Subjects that agree to participate in the extension part of the study, will add on an additional 3 months.

The primary objective of this study is to mechanistically determine the effect of GDMT administered at six months postpartum on GLS at nine months postpartum in African- American patients at high risk due to elevated blood pressures (>120/80 mmHg).

The trial biostatistician will create the randomization schedules using computer-generated random numbers and will have access to treatment group allocation. Below are further details on each arm.

Treatment Arm: Subjects randomized into the treatment arm will be enrolled into the remote patient monitoring program (RPM). Subjects who enroll in the sub-study will utilize the RPM by the University of Chicago Heart Failure Program. This program enables providers to track the number of critical vitals in real time. Patients are equipped and trained to monitor blood pressure, heart rate, weight, temperature, and medication adherence, through a Bluetooth-enabled tablet that integrates and transmits data to the clinic providers and advanced practitioners. This system is currently in use by the heart failure program at the University of Chicago, including hospital-to-home transition care after hospitalization for decompensated heart failure and long-term outpatient management of chronic heart failure, hypertension, atrial fibrillation, and ischemic heart disease. The heart failure team will provide the tablet, blood pressure cuff, weight scale and training at the subjects baseline visit.

Observational Arm: Subjects randomized to this arm will receive the standard of care based upon the American Heart Association (AHA) and American Congress of Obstetricians and Gynecologists (ACOG) guidelines, which include counseling of increased cardiovascular risk, lifestyle modifications, including a healthy diet, exercise, smoking cessation, and risk factor intervention as determined by the primary care physician. They will not be receiving the RPM program equipment.

Follow-up clinic visit approximately 3 months after they have been randomized will be scheduled in both arms. At this visit the study team will;

Perform a Transthoracic echocardiogram (TTE) Obtain Vital signs Physical Exam Adverse Event check Concomitant Medication check Blood draw for laboratory test

In addition, the study team will conduct monthly telephone interviews of all randomized trial participant's for concomitant medications, adverse events/side effects, and study drug compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18 and 45 years of age
2. African American
3. >120/80 BP at the time of their 6-month visit in the PARENT study
4. Diagnosed with preeclampsia
5. Initially presented to University of Chicago Medical Center (UCMC) for a Singleton Gestation Delivery
6. Completed the 6 month visit in the PARENT study

Exclusion Criteria:

1. Those who cannot provide consent
2. patients with preexisting cardiomyopathy, ischemic or valvular heart disease, pulmonary disease, diabetes mellitus, chronic kidney disease, multiple gestations,
3. Unable to operate the RPM tablet device

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with diagnosed pre-eclampsia
Enrollment: 20 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
GLS percentages | 3 Months
  Compare GLS levels as a percentage (%) at 3 months between patients who received RPM program those in the observational group.

SECONDARY OUTCOMES:
Difference in Activin A levels | 3 Months
  Comparing the difference in Activin A levels in subjects at 3 months between patients who received RPM program those in the observational group.
Left Atrial Volume Index | 3 Months
  Comparing the difference between left atrial volume index, from the subjects baseline to 3 month Transthoracic Echocardiogram (TTE)
Deceleration Time | 3 Months
  Comparing the difference between deceleration time from subjects from their baseline to 3 month TTE
Mean Arterial Pressure | 3 Months
  Difference in mean arterial pressure in subjects, from their baseline to 3 month TTE
Ejection Fraction | 3 Months
  Comparing the difference in the ejection fraction percentages, from the subjects baseline to 3 month TEE.
Mitral Annular Motion | 3 months
  Comparing the difference between mitral annular motion, in millimeters (mm), from subjects baseline to 3 month TTE.

CONTACTS AND LOCATIONS:
Overall Officials: Sajid H Shahul, MD PHD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Hospital, Chicago, Illinois, United States